CLINICAL TRIAL: NCT02123901
Title: THE EFFECT OF WALKING MEDITATION TRAINING ON GLYCEMIC CONTROL AND VASCULAR FUNCTION IN PATIENTS WITH TYPE 2 DIABETES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr.Daroonwan Suksom, Faculty of Sports Science, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPSC-1
Record Dates: First submitted 2014-04-18; First posted 2014-04-28 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes
Keywords: Mind and body Exercise; Flow mediated dilation; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Walking meditation & Walking (Experimental)
  Interventions: Other: Walking Meditation; Other: Walking
- Walking meditation & No exercise (Active Comparator)
  Interventions: Other: Walking Meditation; Other: No exercise

INTERVENTIONS:
Other: Walking Meditation — Walking Meditation training program will be based on aerobic walking exercise combined with Buddhist meditation. The subjects will perform walking on the treadmill while concentrated on foot stepping by voiced "Budd" and "Dha" with each foot step that contacted the floor to practice mindfulness while walking. Walking Meditation will be conducted at mild to moderate intensity (50-60% maximum heart rate) and in phase 2 (week 7-12), the training intensity will be increased to moderate intensity (60-70% maximum heart rate). In both phases the training will be performed for 30 minutes, 3 times per week.
  Other Names: Buddhist Walking Meditation
Other: Walking — Walking training program will be based on aerobic walking exercise. The subjects will perform walking on the treadmill and conducted at mild to moderate intensity (50-60% maximum heart rate) and in phase 2 (week 7-12), the training intensity will be increased to moderate intensity (60-70% maximum heart rate). In both phases the training will be performed for 30 minutes, 3 times per week.
  Arms: Walking meditation & Walking
Other: No exercise — Sedentary life style.
  Arms: Walking meditation & No exercise

SUMMARY:
Walking Meditation training would yield more favorable adaptations than walking alone in improving glycemic control and vascular function in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included type 2 diabetes (as defined by the American Diabetes Association), a baseline glycosylated hemoglobin (HbA1c) value of 7-9%, and no previous exercise training in the past 6 months. All participants were free from diabetic nephropathy, diabetic retinopathy, severe diabetic neurophathy, severe cardiovascular and cerebrovascular diseases.

Exclusion Criteria:

* Participants were excluded if they dropped out or completed less than 80% of the training schedule.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycemic control | Baseline, Week 12
  The glycemic control will be quantified using blood samples. Fasting blood glucose, HbA1c, and insulin will be measured with standard procedures at the clinical laboratory (Bria Lab, Bangkok, Thailand).Homeostasis model assessment (HOMA), the parameter for insulin resistance, will be calculated by using equation of [Fasting glucose (mg/dL) × Insulin level (uU/mL) / 405].
Change from baseline in vascular reactivity | baseline, week 12
  Vascular reactivity or brachial artery flow-mediated dilatation (FMD) will be assessed with the ultrasound equipment (CX50, Philips, USA), using the blood occlusion technique on the right forearm. The brachial artery will be imaged above the antecubital fossa in the longitudinal plane. Baseline data will be monitored and the cuff placed around the right forearm will be inflated to 50 mmHg above systolic blood pressure for 5 minutes and then deflated for 5 minutes of recovery. FMD will be calculated from the formula FMD=(D2-D1)x100/D1 when D1 is the brachial artery diameter at baseline, D2 is the maximal post-occlusion brachial artery diameter

SECONDARY OUTCOMES:
Change from baseline in stress indicators | Baseline, Week 12
  * Plasma cortisol will be measured with standard procedures at the certified clinical laboratory (BRIA Lab, Bangkok, Thailand).
  * Heart rate variability (HRV) will be measured using the Heart rate variability analyzer SA-3000P, Medicore Co.,Ltd, Korea
Change from baseline in physical fitness | Baseline, Week 12
  * Body composition will be measured using Body Composition Analyzer (Model ioi 353, Jawon Medical Co. Ltd., Korea).
  * Maximal oxygen consumption (VO2max) will be assessed by Modified Bruce Protocol for treadmill test with Stationary Gas Analyzer (Vmax™ Encore 29 system, Yorba Linda, CA).
  * Lower muscle strength will be measured with back and leg dynamometer.
Change from baseline in Peripheral arterial stiffness | Baseline, Week 12
  Pulse wave velocity measurement will be assessed with MD6 bidirectional transcutaneous Doppler probe (Hokanson, Bellevue, WA, USA). All subjects were monitored with an EKG and PWV measurements in the computer and used as timing markers for PWV identification.
Change from baseline in ankle-brachial index. | Baseline, Week 12
  Ankle-brachial index will be evaluated with a manual MD6 bidirectional transcutaneous Doppler probe (Hokanson, Bellevue, WA, USA) and will be calculated by dividing the highest ankle systolic blood pressure by the highest brachial systolic blood pressure.
Change from baseline in blood chemistry | Baseline, Week 12
  * Interleukin-6 (IL-6) will be measured in plasma samples with the ELISA kit (Human IL-6 high sensitivity ELISA, eBioscience, Austria).
  * Nitric oxide (NO) will be measured in plasma samples with the commercial assay kit (Colorimetric nitric oxide assay kit, PromoKine, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Daroonwan Suksom, Ph.D., Principal Investigator — Faculty of Sports Science, Chulalongkorn University
Locations (1):
- The Primary Health Promoting Hospital, Prapadang, Changwat Samut Prakan, Thailand

REFERENCES:
- [Background] Mitranun W, Deerochanawong C, Tanaka H, Suksom D. Continuous vs interval training on glycemic control and macro- and microvascular reactivity in type 2 diabetic patients. Scand J Med Sci Sports. 2014 Apr;24(2):e69-76. doi: 10.1111/sms.12112. Epub 2013 Sep 17. PMID 24102912
- See also: Related Info — http://www.diabetes.org/